CLINICAL TRIAL: NCT02739997
Title: A Multicenter, Open-label, Noncomparative, Japanese Phase III Study to Assess the Efficacy and Safety of Ceftolozane/Tazobactam (MK-7625A) Used in Combination With Metronidazole in Japanese Patients With Complicated Intra-abdominal Infection.
Brief Title: Study of Ceftolozane/Tazobactam (MK-7625A) in Combination With Metronidazole in Japanese Participants With Complicated Intra-abdominal Infection (MK-7625A-013)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7625A-013; MK-7625A-013 (Other: Merck Registration Number); 163275 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2016-03-30; First posted 2016-04-15 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Intra-abdominal Infection; Complicated Intra-abdominal Infection
MeSH Terms: conditions — Intraabdominal Infections | interventions — ceftolozane; Tazobactam; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MK-7625A + metronidazole (Experimental): MK-7625A 1.5 g (ceftolozane 1 g/tazobactam 0.5 g) plus metronidazole 500 mg administered as an intravenous (IV) infusion every 8 hours for 4 to 14 days. The dose may be reduced to 750 mg (ceftolozane 500 mg/tazobactam 250 mg) for participants with a creatinine clearance (CrCl) of 30-50 mL/min.
  Interventions: Drug: MK-7625A 1.5 g (ceftolozane 1 g/tazobactam 0.5 g); Drug: metronidazole 500 mg

INTERVENTIONS:
Drug: MK-7625A 1.5 g (ceftolozane 1 g/tazobactam 0.5 g) — MK-7625A 1.5 g (ceftolozane 1 g/tazobactam 0.5 g) administered as an intravenous (IV) infusion
Drug: metronidazole 500 mg — metronidazole 500 mg administered as an IV infusion

SUMMARY:
This is a Phase 3, multi-site, non-randomized, open-label study evaluating the safety and efficacy of MK-7625A 1.5 g (ceftolozane 1 g/tazobactam 0.5 g) plus metronidazole 500 mg for the treatment of Complicated Intra-abdominal Infections (cIAI) in Japanese participants. Efficacy will be primarily assessed by clinical response defined as complete resolution or significant improvement in signs and symptoms of the index infection.

ELIGIBILITY:
Inclusion Criteria:

* Has one of the following diagnoses with evidence of intra-peritoneal infection: cholecystitis (including gangrenous cholecystitis) with rupture, perforation, or progression of the infection beyond the gallbladder wall; diverticular disease with perforation or abscess; appendiceal perforation or periappendiceal abscess; acute gastric or duodenal perforation, traumatic perforation of the intestine; peritonitis due to perforated viscus or following a prior operative procedure; or Intra-abdominal abscess (including liver and spleen).
* Has evidence of systemic infection
* Had or has plans to have surgical intervention within 24 hours of the first dose of study drug
* Has radiographic evidence of perforation or abscess if enrolled preoperatively
* Is able to have intra-abdominal specimen taken at baseline for the microbiological assessment
* Female participants of child bearing potential must not be pregnant (negative human chorionic gonadotropin test) or breastfeeding and must agree to use adequate contraception for the duration of the study and up to 35 days after the last dose of study drug
* Male participants must agree to use adequate contraception for the duration of the study and up to 75 days after the last dose of study drug

Exclusion Criteria:

* Has simple appendicitis; abdominal wall abscess; small bowel obstruction or ischemic bowel disease without perforation; spontaneous bacterial peritonitis associated with cirrhosis and chronic ascites; acute suppurative cholangitis; infected necrotizing pancreatitis; pancreatic abscess; infectious mononucleosis; cystic fibrosis; or pelvic infections
* Has complicated intra-abdominal infection managed by staged abdominal repair (STAR) or open abdomen drainage
* Has had acute gastric or duodenal perforation (≤ 24 hours after) or traumatic perforation of the intestine (≤ 12 hours after) operated on after the perforation occurred
* Is expected to be cured by only surgical intervention without use of systemic antibacterial therapy
* Has used systemic antibacterial therapy for intra-abdominal infection for more than 24 hours prior to the first dose of study drug, unless there is a documented treatment failure with such therapy
* Has severe impairment of renal function (estimated CrCl < 30 mL/minute), or requirement for peritoneal dialysis, hemodialysis or hemofiltration, or oliguria (< 20 mL/hour urine output over 24 hours)
* Has a concomitant infection at the time of randomization, which requires non-study systemic antibacterial therapy in addition to study drug with the exception of an antibacterial with Gram-positive activity only (vancomycin, teicoplanin, linezolid and daptomycin)
* Has used any postoperative non-study antibacterial therapy if enrolled preoperatively
* Has used more than 1 dose of non-study antibacterial therapy following surgery if enrolled postoperatively
* Has hepatic disease
* Is unlikely to survive the 4 to 5 week study period
* Has organic brain or spinal cord disease
* Has any rapidly-progressing disease or immediately life-threatening illness
* Has an immunocompromising condition (i.e., AIDS, hematological malignancy, or bone marrow transplantation, or immunosuppressive therapy) or is receiving ≥ 40 mg of prednisone per day administered continuously for > 14 days prior to study start
* Has a history of any moderate or severe hypersensitivity or allergic reaction to any beta-lactam (β-lactam) antibacterial, including cephalosporins, carbapenems, penicillins, or β-lactamase inhibitors, or metronidazole, or nitroimidazole derivatives
* Is receiving or has received disulfiram within 14 days before receiving study drug or who is currently receiving probenecid
* Has participated in any clinical study of an investigational product within 30 days prior to the first dose of study drug
* Has previously participated in any study of ceftolozane or MK-7625A.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-04-08 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2017-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Li Z, Kang Y, Gao H, Zhao Y, Luo D, Wang D, Zhang X, Yu J, Chu G, Cao J, Wang F, Zhao X, Jensen E, Lin G, Chen G. Pooled data from phase 3 clinical trials comparing the clinical activity of ceftolozane/tazobactam versus meropenem for the treatment of complicated intra-abdominal infections. Infect Dis (Lond). 2026 Jan;58(1):40-51. doi: 10.1080/23744235.2025.2544828. Epub 2025 Sep 6. PMID 40913503
- [Derived] Mikamo H, Monden K, Miyasaka Y, Horiuchi T, Fujimoto G, Fukuhara T, Yoshinari T, Rhee EG, Shizuya T. The efficacy and safety of tazobactam/ceftolozane in combination with metronidazole in Japanese patients with complicated intra-abdominal infections. J Infect Chemother. 2019 Feb;25(2):111-116. doi: 10.1016/j.jiac.2018.10.012. Epub 2018 Dec 6. PMID 30528561

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants with complicated intra-abdominal infection (cIAI) were recruited at 37 study sites in Japan.
Groups:
- MK-7625A + Metronidazole: MK-7625A 1.5 g (ceftolozane 1 g + tazobactam 0.5 g) plus metronidazole 500 mg was administered as an IV infusion every 8 hours for 4 to 14 days.
Period: Overall Study
Arm/Group | MK-7625A + Metronidazole
Started | 100
Completed | 98
Not Completed | 2
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | MK-7625A + Metronidazole
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.1 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 100
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Response (Clinical Cure, Clinical Failure, or Indeterminate) at Test of Cure (TOC)
Description: The percentage of participants with clinical responses (cure, failure, or indeterminate) at TOC was determined. Clinical cure was defined as "complete resolution or significant improvement in signs and symptoms of the index infection, such that no additional antibacterial therapy or surgical or drainage procedure is required". Clinical failure was defined as "death related to IAI at any time point; persisting or recurrent infection within the abdomen requiring additional intervention to cure; need for treatment with additional antibiotics for ongoing IAI symptoms; or post-surgical wound infection that requires additional antimicrobial therapy and/or non-routing wound care". Indeterminate was defined as "study data are not available for evaluation for any reason, including death during the study period unrelated to the index infection; or extenuating circumstances that preclude classification as cure or failure".
Time Frame: Day 28 (28 days after initiating study therapy)
Population: Clinically evaluable participants were defined as those who received study therapy for ≥3 days, had 80-120% study therapy compliance, met criteria for cIAI, adhered to study procedures, and had a clinical response at the TOC visit within the specified visit window are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-7625A + Metronidazole
Number analyzed (Participants) | 88
Percentage of Participants
  Success | 92.0
  Failure | 8.0
  Indeterminate | 0.0

2. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: The percentage of participants with ≥1 AEs was determined. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to Day 42 (up to 28 days after completing study therapy)
Population: All participants who received ≥1 dose of study therapy are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MK-7625A + Metronidazole
Number analyzed (Participants) | 100
Percentage of Participants | 62.0 [51.7 to 71.5]

3. Primary Outcome: Percentage of Participants Discontinuing Study Drug Due to AEs
Description: The percentage of participants withdrawing from study therapy due to an AE was determined.
Time Frame: Up to Day 14
Population: All participants who received ≥1 dose of study therapy are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MK-7625A + Metronidazole
Number analyzed (Participants) | 100
Percentage of Participants | 0.0 [0.0 to 3.6]

4. Secondary Outcome: Percentage of Participants With Clinical Response (Clinical Cure, Clinical Failure, or Indeterminate) at End Of Therapy (EOT)
Description: The percentage of participants with clinical responses (cure, failure, or indeterminate) at EOT was determined. Clinical cure was defined as "complete resolution or significant improvement in signs and symptoms of the index infection, such that no additional antibacterial therapy or surgical or drainage procedure is required". Clinical failure was defined as "death related to IAI at any time point; persisting or recurrent infection within the abdomen requiring additional intervention to cure; need for treatment with additional antibiotics for ongoing IAI symptoms; or post-surgical wound infection that requires additional antimicrobial therapy and/or non-routing wound care". Indeterminate was defined as "study data are not available for evaluation for any reason, including death during the study period unrelated to the index infection; or extenuating circumstances that preclude classification as cure or failure".
Time Frame: Up to Day 14
Population: Clinically evaluable participants were defined as those who received study therapy for ≥3 days, had 80-120% study therapy compliance, met criteria for cIAI, adhered to study procedures, and had a clinical response at EOT visit within the specified visit window are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-7625A + Metronidazole
Number analyzed (Participants) | 92
Percentage of Participants
  Success | 94.6
  Failure | 5.4
  Indeterminate | 0.0

5. Secondary Outcome: Percentage of Participants With Clinical Response (Clinical Cure, Clinical Failure, or Indeterminate) at Late Follow-Up (LFU)
Description: The percentage of participants with clinical responses (cure, failure, or indeterminate) at LFU was determined. Clinical cure was defined as "complete resolution or significant improvement in signs and symptoms of the index infection, such that no additional antibacterial therapy or surgical or drainage procedure is required". Clinical failure was defined as "death related to IAI at any time point; persisting or recurrent infection within the abdomen requiring additional intervention to cure; need for treatment with additional antibiotics for ongoing IAI symptoms; or post-surgical wound infection that requires additional antimicrobial therapy and/or non-routing wound care". Indeterminate was defined as "study data are not available for evaluation for any reason, including death during the study period unrelated to the index infection; or extenuating circumstances that preclude classification as cure or failure".
Time Frame: Up to Day 42 (28 days after completing study therapy)
Population: Clinically evaluable participants were defined as those who received study therapy for ≥3 days, had 80-120% study therapy compliance, met criteria for cIAI, adhered to study procedures, and had a clinical response at LFU visit within the specified visit window are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-7625A + Metronidazole
Number analyzed (Participants) | 85
Percentage of Participants
  Success | 90.6
  Failure | 9.4
  Indeterminate | 0.0

6. Secondary Outcome: Percentage of Participants With Microbiological Response (Eradication, Persistence, or Indeterminate) at EOT
Description: The percentage of participants with microbiological responses (eradication, persistence, or indeterminate) at EOT was determined. Eradication was defined as "absence of the baseline pathogen in a specimen". Persistence was defined as "presence of the baseline pathogen in a specimen". Indeterminate was defined as "Baseline culture either not obtained or has an assessment of no growth, or any other circumstance that makes it impossible to define the microbiological response".
Time Frame: Up to Day 14
Population: Expanded microbiologically evaluable participants were defined as those who received study therapy for ≥3 days, had 80-120% study therapy compliance, met criteria for cIAI, adhered to study procedures, had a microbiological response at the EOT visit within the specified visit window, and have ≥1 identified intra-abdominal pathogen are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-7625A + Metronidazole
Number analyzed (Participants) | 65
Percentage of Participants
  Eradication | 93.8
  Persistence | 6.2
  Indeterminate | 0.0

7. Secondary Outcome: Percentage of Participants With Microbiological Response (Eradication, Persistence, or Indeterminate) at TOC
Description: The percentage of participants with microbiological response (eradication, persistence, or indeterminate) at TOC was determined. Eradication was defined as "absence of the baseline pathogen in a specimen". Persistence was defined as "presence of the baseline pathogen in a specimen". Indeterminate was defined as "Baseline culture either not obtained or has an assessment of no growth, or any other circumstance that makes it impossible to define the microbiological response".
Time Frame: Day 28 (28 days after initiating study therapy)
Population: Expanded microbiologically evaluable participants were defined as those who received study therapy for ≥3 days, had 80-120% study therapy compliance, met criteria for cIAI, adhered to study procedures, had a microbiological response at the TOC visit within the specified visit window, and have ≥1 identified intra-abdominal pathogen are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-7625A + Metronidazole
Number analyzed (Participants) | 61
Percentage of Participants
  Eradication | 90.2
  Persistence | 9.8
  Indeterminate | 0.0

8. Secondary Outcome: Percentage of Participants With Microbiological Response (Eradication, Persistence, or Indeterminate) by Pathogen at EOT
Description: The percentage of participants with per-pathogen microbiological responses at EOT was determined. Individual pathogens were identified at baseline, and the overall percentage of participants with eradication or presumed eradication within each pathogen category are shown.
Time Frame: Up to Day 14
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MK-7625A + Metronidazole
Number analyzed (Participants) | 65
Percentage of Participants
  Gram-Negative Aerobes: number analyzed (Participants) | 55
  Gram-Negative Aerobes | 94.5 [84.9 to 98.9]
  Gram-Positive Aerobes: number analyzed (Participants) | 40
  Gram-Positive Aerobes | 95.0 [83.1 to 99.4]
  Gram-Negative Anaerobes: number analyzed (Participants) | 44
  Gram-Negative Anaerobes | 97.7 [88.0 to 99.9]
  Gram-Positive Anaerobes: number analyzed (Participants) | 21
  Gram-Positive Anaerobes | 90.5 [69.6 to 98.8]

9. Secondary Outcome: Percentage of Participants With Microbiological Response (Eradication, Persistence, or Indeterminate) by Pathogen at TOC
Description: The percentage of participants with per-pathogen microbiological responses at TOC was determined. Individual pathogens were identified at baseline, and the overall percentage of participants with eradication or presumed eradication within each pathogen category are shown.
Time Frame: Day 28 (28 days after initiating study therapy)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MK-7625A + Metronidazole
Number analyzed (Participants) | 61
Percentage of Participants
  Gram-Negative Aerobes: number analyzed (Participants) | 53
  Gram-Negative Aerobes | 90.6 [79.3 to 96.9]
  Gram-Positive Aerobes: number analyzed (Participants) | 38
  Gram-Positive Aerobes | 89.5 [75.2 to 97.1]
  Gram-Negative Anaerobes: number analyzed (Participants) | 42
  Gram-Negative Anaerobes | 95.2 [83.8 to 99.4]
  Gram-Positive Anaerobes: number analyzed (Participants) | 20
  Gram-Positive Anaerobes | 85.0 [62.1 to 96.8]

ADVERSE EVENTS:
Time Frame: Up to Day 42
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. All participants who received ≥1 dose of study drug are included.
Arm/Group | MK-7625A + Metronidazole
All-Cause Mortality (participants affected / at risk) | 1/100
Serious Adverse Events (participants affected / at risk) | 10/100
Other Adverse Events (participants affected / at risk) | 32/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-7625A + Metronidazole (N=100)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Eating disorder (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-7625A + Metronidazole (N=100)
Constipation (Gastrointestinal disorders) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 7 (7)
Alanine aminotransferase increased (Investigations) | 11 (11)
Aspartate aminotransferase increased (Investigations) | 13 (13)
Insomnia (Psychiatric disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-21): https://cdn.clinicaltrials.gov/large-docs/97/NCT02739997/Prot_SAP_000.pdf